#### Corporate Clinical Development Template CCD-6230.T01 Revision 01



#### Statistical Analysis Plan

| Protocol Number/version | MPS-17IPVSS02/Version 2.0 - 06 May 2019 (Amendment 1) |
|---|---|
| Protocol Title | A Randomized, Single-Center, Partially Blinded, Evaluation of the Time- |
| | Dependent Antimicrobial Effectiveness of Swabsticks Impregnated with 2% |
| | (w/v) Chlorhexidine Gluconate in 70% (v/v) Isopropyl Alcohol in Healthy Vol- |
| | unteers |
| SAP Date | August 2, 2019 |

| Version History | Action |
|-----------------|------------------|
| August 2, 2019 | Original Release |

This report is proprietary to Becton Dickinson. No part of it may be distributed or shared with persons other than BD associates without written permission from Global Clinical Development (GCD).

### Approval

| Function | Name | Signature |
|---|---|---|
| Statistician (Author) | | $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ |
| Study Manager | | This document is signed electronically in the eTMF system. |
| Associate Director, Statistics | | This document is signed electronically in the eTMF system. |

NCT Number: [NCT04035161] (Number added post-approval per CT.gov requirement)

# Contents

| 1 | List | of Abbreviations and Definitions | 5 |
|---|---|---|---|
| 2 | Ove | erall Study Description | 6 |
| | 2.1 | Study Background | 6 |
| | 2.2 | Objectives | 6 |
| | | 2.2.1 Safety Objectives | 6 |
| | | 2.2.2 HC Objectives | 6 |
| | | 2.2.2.1 Primary Efficacy Objectives | 6 |
| | | 2.2.2.2 Exploratory Objective | 6 |
| | | 2.2.3 FDA Objectives | 7 |
| | | 2.2.3.1 Primary Objectives | 7 |
| | | 2.2.3.2 Secondary Objectives | 7 |
| | | 2.2.3.3 Exploratory Objectives | 7 |
| | 2.3 | Study Design | 7 |
| | 2.4 | Endpoints | 9 |
| | 2.5 | Acceptance Criteria | 9 |
| | | Treespecial Critical | |
| 3 | San | nple Size | 11 |
| | 3.1 | HC Analysis | 11 |
| | 3.2 | | 11 |
| 4 | Inte | ended Statistical Software | 11 |
| 5 | Dat | $z_{\mathbf{a}}$ | <b>12</b> |
| | 5.1 | Database Information | 12 |
| | 5.2 | Data Sets Analyzed | 12 |
| | 5.3 | Protocol Deviations and Use of Associated Data | 12 |
| | 5.4 | Analysis Population $Set(s)$ | 12 |
| • | Cu. | | - 1 |
| 6 | | | 14 |
| | 6.1 | | 14 |
| | | 6.1.1 $Log_{10}$ CFU/cm <sup>2</sup> of skin | 14 |
| | | 6.1.2 Log Reduction | 14 |
| | | 6.1.3 Responder Rate | 14 |
| | | 6.1.4 Product Weight | 15 |
| | 6.2 | Analysis Methods | 15 |
| | | 6.2.1 HC Analysis | 15 |
| | | 6.2.1.1 Summary Statistics | 15 |
| | | 6.2.1.2 Primary Analysis | 15 |
| | | 6.2.1.3 Exploratory Analysis | 15 |
| | | 6.2.2 FDA Analysis | 16 |
| | | 6.2.2.1 Summary Statistics | 16 |
| | | 6.2.2.2 Primary Analysis | 16 |
| | | 6.2.2.3 Secondary Analysis | 16 |
| | | 6.2.3 Safety Analysis | 17 |
| | 6.3 | Adjustments for Multiple Objectives | 18 |

| | 6.4 Handling of Missing Data and Sensitivity Analysis | 18<br>19 |
|---|---|---|
| | 6.5 Demographics/Other Descriptive Information | 20 |
| 7 | References | 21 |
| 8 | Appendix | 22 |
| A | Tables | 22 |
| | A.1 Analysis Population Set(s) | 22 |
| | A.2 HC Analysis | 23 |
| | A.3 FDA Analysis | $\frac{25}{27}$ |
| | A.5 Sensitivity Analysis | 29 |
| | A.6 Demographics | 31 |
| В | Listings | 32 |
| $\mathbf{C}$ | Figures | 35 |
| | C.1 HC Analysis | 35 |
| | C.2 FDA Analysis | 36 |
| $\mathbf{T}$ | ables and Listings | |
| | 1 mITT Data Set for Each Anatomical Site and Expected Minimum Efficacy Standards | 1( |
| | 2 Parameters Used in Sample Size Calculations For HC Analysis | 11 |
| | 3 Parameters Used in Sample Size Calculations For FDA Analysis | 11 |
| | Guideline on Use of Associated Data in Analysis for Potential Protocol Deviations | 13 |
| | A.1.1 Overall Subject Disposition | $\frac{22}{22}$ |
| | A.1.3 Number of Evaluable Subjects for FDA Analysis | $\frac{22}{22}$ |
| | A.2.1 mITT/PP - Summary Statistics for HC Analysis - Log CFU | 23 |
| | A.2.2 mITT/PP - Summary Statistics for HC Analysis - Log Reduction | 23 |
| | A.2.3 mITT/PP - Summary Statistics for HC Analysis - Product Weight | 23 |
| | A.2.4 mITT/PP - Analysis Results for HC Analysis - Log Reduction at 30 Seconds and 6 | 0.0 |
| | Hours | 23 |
| | A.2.5 mITT/PP - Analysis Results for for HC Analysis - Log Reduction at 10 Minutes A.2.6 mITT/PP - Analysis Results for for HC Analysis - Difference in Log Reduction | $\frac{24}{24}$ |
| | A.3.1 mITT/PP - Summary Statistics for FDA Analysis - Log CFU | $\frac{24}{25}$ |
| | A.3.2 mITT/PP - Summary Statistics for FDA Analysis - Log Reduction | 25 |
| | A.3.3 mITT/PP - Summary Statistics for FDA Analysis - Responder Rate at 6 Hours | 25 |
| | A.3.4 mITT/PP - Summary Statistics for FDA Analysis - Product Weight | 25 |
| | A.3.5 mITT/PP - Analysis Results for FDA Analysis - ATE at 10 Minutes | 26 |

| Α | 3.0 | mITT/PP - Analysis Results for FDA Analysis - ATE at 30 Seconds | 26 |
|---|---|---|---|
| A | .4.1 | ITT - Summary Statistics for Irritation Scores for Abdomen/Groin at Baseline/30 | |
| | | Seconds/10 Minutes/6 Hours | 27 |
| A | .4.2 | ITT - Adverse Events Summary | 27 |
| A | 4.3 | ITT - Safety Analysis - Overall Comparisons for Erythema/Edema/Rash/Dryness | 28 |
| A | .4.4 | ITT - Safety Analysis - Subgroup Comparisons for Irritation Scores | 28 |
| A | 5.1 | Pooled Analysis Results Based on Imputated Datasets for HC Objectives - Log Reduction | 29 |
| A | 5.2 | Pooled Analysis Results Based on Imputated Datasets for FDA Objectives - ATE | 29 |
| A | 5.3 | Tipping Point Analysis for HC Objectives - Log Reduction | 29 |
| A | 5.4 | Tipping Point Analysis for FDA Objectives - ATE | 30 |
| A | 5.5 | Sensitivity Analysis for FDA Objectives - Responder Rate at 6 Hours | 30 |
| A | .6.1 | ITT - Demographics | 31 |
| В | .1 | Protocol Deviations | 32 |
| В | .2 | Subjects with Excluded Data for HC Analysis | 32 |
| В | .3 | Subjects with Excluded Data for FDA Analysis | 32 |
| В | .4 | Subjects who Did Not Complete the Study | 32 |
| В | .5 | Subjects Not Passing Treatment-day Baseline Criteria | 33 |
| В | .6 | Adverse Events | 33 |
| В | .7 | Serious Adverse Events | 33 |
| В | .8 | Procedure Overview - Sampling Fluid | 33 |
| В | .9 | Procedure Overview - Dressing Application | 34 |
| В | .10 | Core Lab Procedure Overview - Sample Solution | 34 |
| В | .11 | Product Failures/Lab Accidents/User Errors | 34 |
| Fig | ure | es | |
| | | mITT/PP - Log Reduction with 95% CI (Example Data Only) | 35 |
| C | .2.1 | mITT/PP - ATE with 95% CI (Example Data Only) | 36 |



#### 1 List of Abbreviations and Definitions

- AC: Active Control
- **AE:** Adverse Event
- ANOVA: Analysis of Variance
- ASTM: American Society for Testing and Materials
- ATE: Average Treatment Effect
- BD: Becton Dickinson and Company
- **CFU:** Colony Forming Units
- CHG: Chlorhexidine Gluconate
- CI: Confidence Interval
- CRF: Case Report/Record Form
- EDC: Electronic Data Capture
- FDA: Food and Drug Administration
- GCD: Global Clinical Development
- HC: Health Canada
- IP: Investigational Product
- ITT: Intent to Treat
- MAR: Missing at Random
- mITT: Modified Intent to Treat
- NC: Negative Control
- **PP:** Per-Protocol
- RS: Reference Standard
- SAE: Serious Adverse Event
- **SD**: Standard Deviation



### 2 Overall Study Description

### 2.1 Study Background

In this study, the antimicrobial activity of the investigational product (IP), a single Swabstick impregnated with 1.75 mL of 2% (w/v) chlorhexidine gluconate (CHG) in 70% (v/v) isopropyl alcohol, will be investigated according to established testing requirements described by Health Canada (HC) and the US FDA.

For evaluation of antimicrobial activity using the HC analysis criteria, immediate antimicrobial activity will be evaluated at 30 seconds and persistent antimicrobial activity will be evaluated at 6 hours post-product application on the abdomen and the groin for the IP. A reference standard, 60% v/v 1-Propanol, will be applied with a single Swabstick and will also be compared to the same log reduction standards as the IP.

For evaluation of antimicrobial activity using the FDA analysis criteria, the immediate antimicrobial activity will be evaluated at 10 minutes post-product application on the abdomen and the groin (primary objectives) and at 30 seconds post-product application on the abdomen only (secondary objectives). Persistent antimicrobial activity will be evaluated at 6 hours post-product application on the abdomen and the groin.

#### 2.2 Objectives

#### 2.2.1 Safety Objectives

To evaluate safety using skin irritation scores and the incidence of adverse events reported during the study for all study products.

#### 2.2.2 HC Objectives

#### 2.2.2.1 Primary Efficacy Objectives

To demonstrate the immediate and persistent antimicrobial activity of a single Swabstick impregnated with 2% (w/v) chlorhexidine gluconate in 70% (v/v) isopropyl alcohol at 30 seconds and 6 hours post-product application.

The reference standard of 60% v/v 1-propanol (RS) applied with a Swabstick, should meet the same efficacy standards described in Table 1 as the IP.

#### 2.2.2.2 Exploratory Objective

- To evaluate the  $\log_{10}$  CFU/cm<sup>2</sup> reductions from baseline for the IP and RS at each anatomical site, abdomen and groin, at 10 minutes post-product application.
- To determine if the 30-second, 10 minutes and 6 hour  $\log_{10}$  CFU/cm<sup>2</sup> reductions on the abdomen and groin for the IP are not statistically worse than those for 60% v/v 1-propanol post-product application.



#### 2.2.3 FDA Objectives

#### 2.2.3.1 Primary Objectives

To demonstrate the immediate and persistent antimicrobial properties of a single Swabstick impregnated with 2% (w/v) chlorhexidine gluconate in 70% (v/v) isopropyl alcohol to ChloraPrep SEPP Clear Applicator AC and a NC of 0.9% normal saline at 10 minutes and 6 hours post product application.

- To demonstrate immediate antimicrobial efficacy at 10 minutes post-application (four co-primary objectives):
  - To demonstrate the non-inferiority of the average treatment effect (ATE) of the IP compared to the AC on the abdomen.
  - To demonstrate the non-inferiority of the average treatment effect (ATE) of the IP compared to the AC on the groin.
  - To demonstrate the superiority of the ATE of the IP compared to the NC on the abdomen.
  - To demonstrate the superiority of the ATE of the IP compared to the NC on the groin.
- To evaluate persistent antimicrobial efficacy at 6 hours post-product application. Log<sub>10</sub> bacterial counts for each product application site will be converted to a binary (yes or no) success measure with success defined as having skin flora counts that are less than or equal to the baseline skin flora counts. Responder rates at 6 hours post-product application will be summarized descriptively for each product on each body site.

#### 2.2.3.2 Secondary Objectives

To demonstrate antimicrobial efficacy at 30 seconds post-application (two secondary objectives):

- To demonstrate the non-inferiority of the average treatment effect (ATE) of the IP compared to the AC on the abdomen.
- To demonstrate the superiority of the ATE of the IP compared to the NC on the abdomen.

These two secondary objectives will be evaluated only when the four co-primary efficacy objectives pass both non-inferiority and superiority criteria. The secondary objectives will declare success when and only when all four primary and two secondary objectives pass both non-inferiority and superiority criteria.

#### 2.2.3.3 Exploratory Objectives

- To evaluate the  $\log_{10}$  CFU/cm<sup>2</sup> reductions from baseline for the IP, AC, and NC at each anatomical site at 30 seconds, 10 minutes and 6 hours.
- To calculate the product weight expression from product application [i.e., product weight prior to product application (g) product weight post-product application (g)].

#### 2.3 Study Design

This single site study is a randomized, controlled, partially blinded, design enrolling a minimum of 516 healthy volunteers, where each subject will receive two of the planned study products on the product application sites of the abdomen and/or groin. In this study, the antimicrobial activity of the investigational product (IP), a single Swabstick impregnated with 1.75 mL of 2% (w/v) chlorhexidine gluconate (CHG) in 70% (v/v) isopropyl alcohol, will be investigated according to established testing



requirements described by Health Canada (HC) and the US FDA. The study methods for this evaluation will be based on ASTM Standard Test Method E1173-15 [1].

Descriptions of study products are shown below.

- Investigational Product (IP): Single Swabstick impregnated with 2% (w/v) chlorhexidine gluconate (CHG) in 70% (v/v) isopropyl alcohol
- Reference Standard (RS): 60% (v/v) 1-propanol applied with a single Swabstick
- Active Control (AC): Chlora Prep SEPP - 2% chlorhexidine gluconate in 70% (v/v) isopropyl alcohol
- Negative Control (NC): 0.9% normal saline applied with a single Swabstick

A minimum of 516 evaluable subjects will be required to achieve a minimum of 192 evaluable product application sites for groin and abdominal regions for 60% (v/v) 1-propanol (RS) and 280 evaluable product application sites for groin and abdominal regions for each of the other three study product arms.

Due to the imbalance of the sample size between RS and other products, RS cannot be blinded and is coded as B and all the other three products will be blinded with assigned study product codes A, C, or D. More information about blinding and methods to reduce bias may be found in the protocol for this study.

The effectiveness of the neutralizer system must be validated prior to the main treatment study start date to demonstrate that the antimicrobials are effectively neutralized and there is no effect on the growth of microorganisms. GCD statistics group will not perform any summary or analysis for the neutralization validation data so this statistical analysis plan (SAP) only applies to the main treatment study.



#### 2.4 Endpoints

- Safety Endpoints: Skin reactions using the modified Berger Bowman irritation assessment scale and the incidence of AEs reported during the study.
- Efficacy Endpoints: Log<sub>10</sub> CFU/cm<sup>2</sup> of resident microbes on skin before and after each product application at 30 seconds, 10 minutes and 6 hours on the abdomen and groin.
- Exploratory Endpoints: Product weight prior to product application (g) and post-product application (g) on the abdomen and groin.

#### 2.5 Acceptance Criteria

To be included in the primary analysis [modified intent-to-treat (mITT) data set], a product application site must have a Product Application Day microbial baseline within the stated requirements. Table 1 summarizes the baseline criteria for the mITT data set for each anatomical site and the expected minimum efficacy country specific standards.

For HC primary objectives, it will declare success when and only when all four primary objectives pass HC analysis acceptance criteria.

For FDA primary objectives [10-minute (abdomen and groin) post-product application time point], it will declare success when and only when all four primary objectives pass FDA analysis acceptance criteria. For FDA secondary objectives [30-second (abdomen only) post-product application time point], a gatekeeping procedure will be applied: the efficacy analysis for two secondary objectives will be performed only when all four primary objectives [10-minute (abdomen and groin) post-product application time point] pass the acceptance criteria and it will declare success when and only when all four primary and two secondary objectives pass FDA analysis acceptance criteria.

For responder rate at 6 hours, no acceptance criteria are applied.

Table 1: mITT Data Set for Each Anatomical Site and Expected Minimum Efficacy Standards

| Anatomical | Product | HC Analysis | HC Analysis | FDA Analysis | FDA Analysis |
|---|---|---|---|---|---|
| Product | Application | Acceptance | Acceptance | Acceptance | Acceptance |
| Application | Day Baseline | Criteria at 30 | Criteria at 6 Hours, | Criteria at 30 | Criteria at 10 |
| Site | Criteria | Seconds, Primary | Primary Objectives | Seconds, Secondary | Minutes, Primary |
| | | Objectives | | Objectives | Objectives |
| Abdomen | 3.20 to 6.00 | Immediate | Persistence | At 30 seconds the | At 10 minutes the |
| | $\log_{10}$ | effectiveness for the IP | effectiveness for the IP | upper two-sided 95% | upper two-sided $95\%$ |
| | $\mathrm{CFU/cm^2}$ | is at least a $2-\log_{10}$ | is at least a $2-\log_{10}$ | confidence bound of | confidence bound of |
| | | CFU/cm <sup>2</sup> reduction | CFU/cm <sup>2</sup> reduction | the average treatment | the average treatment |
| | | from baseline skin | from baseline skin. | effect (ATE) of IP - | effect (ATE) of $IP$ - |
| | | flora counts at 30 | flora counts at 6 | AC should be less | AC should be less |
| | | seconds. | hours. | than $0.5 \log_{10}$ . At 30 | than $0.5 \log_{10}$ . At 10 |
| | | | | seconds the lower | minutes the lower |
| | | | | two-sided $95\%$ | two-sided $95\%$ |
| | | | | confidence bound of | confidence bound of |
| | | | | the ATE of NC - IP | the ATE of NC - IP |
| | | | | should be greater than | should be greater than |
| | | | | $1.2 \log_{10}$ . | $1.2 \log_{10}$ . |
| Groin | 5.50 to 7.50 | Immediate | Persistence | None | At 10 minutes the |
| | $\log_{10}$ | effectiveness for the IP | effectiveness for the IP | | upper two-sided $95\%$ |
| | $\mathrm{CFU/cm^2}$ | is at least a $3-\log_{10}$ | is at least a $3-\log_{10}$ | | confidence bound of |
| | | CFU/cm <sup>2</sup> reduction | CFU/cm <sup>2</sup> reduction | | the average treatment |
| | | from baseline skin | from baseline skin. | | effect (ATE) of IP - |
| | | flora counts at 30 | flora counts at 6 | | AC should be less |
| | | seconds. | hours. | | than $0.5 \log_{10}$ . At 10 |
| | | | | | minutes the lower |
| | | | | | two-sided $95\%$ |
| | | | | | confidence bound of |
| | | | | | the ATE of NC - IP |
| | | | | | should be greater than |
| | | | | | $1.2 \log_{10}$ . |





### 3 Sample Size

### 3.1 HC Analysis

To evaluate the primary efficacy objective for HC analysis a sample size of at least 192 evaluable sites per study product arm (IP or RS) per body site can achieve > 95% power to pass HC analysis acceptance criteria for all four objectives (IP only) using one-sample t-test (two-sided), with the following assumptions in Table 2.

Two-sided test Type I error  $(\alpha)$ : 0.05 Time Point Study Standard Standard Log Reduction: Log Reduction: Product Deviation for Log Deviation for Log Abdomen  $(\log_{10})$ Groin  $(\log_{10})$ Reduction: Reduction: Groin Abdomen 30 seconds ΙP 1.14 1.43 3.47 3.38 6 hours ΙP 1.22 1.24 3.43 3.50

Table 2: Parameters Used in Sample Size Calculations For HC Analysis

#### 3.2 FDA Analysis

To evaluate the primary and secondary objectives for the US FDA analysis a sample size of 280 evaluable sites per study product arm (IP, AC or NC) per body site can achieve > 95% power to demonstrate the non-inferiority of the Investigational Product (IP) as compared to the Active Control (AC) and the superiority of the IP as compared to the negative control (NC) in antimicrobial effect at 30-second (abdomen only) and 10-minute (abdomen and groin) post-product application time point for all six objectives, with the following assumptions in Table 3.

| and of I diameters of the Sample Size Calculations for I Diff I many |
|---|
| Two-sided test Type I error $(\alpha): 0.05$ |
| Average Treatment Effect Abdomen $(\log_{10})$ Groin $(\log_{10})$ |
| IP - AC 0.06 0.10 |
| NC - IP 1.58 2.31 |
| Standard deviation for each product on Abdomen: $1.05 \log_{10}$ |
| Standard deviation for each product on Groin: 1.2 log <sub>10</sub> |

Table 3: Parameters Used in Sample Size Calculations For FDA Analysis

The overall power to pass both HC analysis and FDA analysis acceptance criteria is > 90%.

#### 4 Intended Statistical Software

The analyses will be performed using R version 3.6.0 (2019-04-26) [2] or higher. R libraries and versions that are used for analyses will be listed.



#### 5 Data

#### 5.1 Database Information

Data will be captured by electronic case report forms (eCRFs) and provided to study statistician and statistical programmer by Data Management. More information on database management may be found in Data Management Plan for this study.

#### 5.2 Data Sets Analyzed

- The full intent-to-treat (ITT) data set (all randomized subjects that received study product) will be used for the safety analysis.
- A modified intent-to-treat (mITT) data set will be used for efficacy analyses. Inclusion for the mITT data set is evaluated for each anatomical site (left and right for the groin and abdomen). For each anatomical site, product application day baseline criteria must be met (refer to Table 1 for product application day baseline criteria) in order to be included in the mITT data set.
- Analyses conducted on the mITT data set will also be conducted on the Per Protocol data set
  as supportive analyses when Per Protocol data are different from mITT data. The Per-Protocol
  data set will include evaluable product application sites from the mITT data set that adhere to
  defined assessments and procedures in the protocol central to patient enrollment, safety, rights
  or wellbeing, as well as the completeness, accuracy and reliability of study data.

#### 5.3 Protocol Deviations and Use of Associated Data

Table 4 lists pre-defined potential protocol deviations and rules for use of associated data in analysis, which has been documented in a note-to-file "MPS-17IPVSS02\_Guideline\_Protocol\_Deviations\_Data\_Use.pdf". For any additional protocol deviations or issues that are not listed in Table 4, exclusion of the data from each population set will be reviewed and finalized on a case by case prior to the database lock.

All protocol deviations for this study will be listed (cf. Listing B.1). Any data that are excluded from any analysis will be listed indicating from which population sets data are excluded (cf. Listings B.2 for HC analysis and B.3 for FDA analysis).

#### 5.4 Analysis Population Set(s)

For subject disposition, refer to Table A.1.1. Subjects who did not complete the study will be listed along with the status at the end of study (cf. Listing B.4).

For each analysis (HC analysis and FDA analysis), the number of subjects evaluable for ITT (randomized and treated/study product received), mITT and per-protocol (PP) analyses for CFU count and product weight per body site/location will be tabulated (cf. Tables A.1.2 for HC analysis and A.1.3 for FDA analysis). Subjects who were randomized and treated but did not pass the product application day baseline criteria (not eligible for mITT or PP analysis) will be listed (cf. Listing B.5).



Table 4: Guideline on Use of Associated Data in Analysis for Potential Protocol Deviations

| | | Use of | Associated | Data in A | Analysis |
|---|---|---|---|---|---|
| Category | $egin{aligned} ext{Description of Deviation} \ ext{(Examples)} \end{aligned}$ | mITT<br>CFU<br>count | PP<br>CFU<br>count | mITT<br>weight | PP<br>weight |
| Randomization<br>error | Incorrect product applied based on<br>randomization schedule or Subject<br>received application of one or more<br>incorrect products (grouped based on<br>product applied) | Yes | No | Yes | No |
| | Subject received correct product but product was applied to incorrect side of the body based on randomization schedule Sample taken from incorrect sample site within the treatment area based on randomization schedule | | | | |
| Deviation from defined procedure | Loss of partial sampling volume | Yes | No | Yes | No |
| | Samples not plated in the 30 minute timeframe from collection Subject leaves the study site but returns for assessments Product application time outside of $30 \text{ seconds} \pm 5 \text{ seconds}$ on the abdomen or $2 \text{ minutes} \pm 5 \text{ seconds}$ on the groin | | | | |
| Clinical<br>assessment not<br>done | Plates not dosed or plates contamination | No | No | No | No |
| Clinical<br>assessment<br>outside of window | Sampling time outside specified windows | Yes | No | Yes | No |
| Other | Pooling of samples from different<br>subjects or different time points from<br>the same subject | No | No | No | No |
| | Product weight error (difference in weights between pre application and post application less than 0 or greater than 2 grams) | Yes | Yes | No | No |



### 6 Statistical Analysis/Calculations

#### 6.1 Derived Variables

### $6.1.1 \quad \text{Log}_{10} \text{ CFU/cm}^2 \text{ of skin}$

Raw colony counts from each dilution will be recorded on the appropriate eCRFs for each subject. The average number of microorganisms recovered will be calculated using the formula below to convert the bacterial counts into  $\log_{10}$  CFU/cm<sup>2</sup> of skin:

$$R = log_{10} \left\lceil \frac{F\left(\frac{\sum_{i=1}^{3} C_{i}}{n}\right) D}{A} \right\rceil \tag{1}$$

Where:

R= the average CFU count in  $\log_{10}$  scale per cm $^2$  of skin.

F = Total number of mL of stripping fluid added to the sampling cylinder (6 mL). Note: If sample solution is lost during the procedure for a certain time point, the F value for that time point will change from 6 mL to the "Volume Remaining (mL)" recorded in the Core Lab Procedure Overview eCRFs.

 $\frac{\sum_{i=1}^{3} C_i}{n}$  = average of the triplicate colony counts used for each sample collected (n = 3).

D = Dilution factor of the plates counted. One of  $10^0$ ,  $10^1$ ,  $10^2$ ,  $10^3$ ,  $10^4$ , or  $10^5$ .

A = Inside area of the sampling cylinder in cm<sup>2</sup> (3.80 cm<sup>2</sup>).

The average CFU/mL, CFU/cm<sup>2</sup>, and  $\log_{10}$  CFU/cm<sup>2</sup> will be calculated for samples from each product application site in the same manner.

In order to avoid potential calculation problems due to taking the logarithm of zero, values of less than  $1 \text{ CFU/cm}^2$  will be treated as  $1 \text{ CFU/cm}^2$ , such that the  $\log_{10}$  transformation is not less than zero.

If colonies on one of the plates are uncountable, the average count from the remaining plates will be used. If colonies on two of the plates are uncountable, the count from the remaining plate will be used. If colonies on three plates are all uncountable, the average count will be missing.

#### 6.1.2 Log Reduction

 $Log_{10}$  CFU/cm<sup>2</sup> reductions from baseline will be calculated separately for each subject, each of the four sites (left and right for the abdomen and groin), and each post-product application sampling time by taking the baseline  $log_{10}$  CFU/cm<sup>2</sup> values and then subtracting the  $log_{10}$  CFU/cm<sup>2</sup> values for the samples taken after baseline. The mean  $log_{10}$  CFU/cm<sup>2</sup> changes from baseline will be calculated separately for each product, at each anatomical site (abdomen and groin), and at each post-product application sampling time point (30 seconds, 10 minutes and 6 hours).

#### 6.1.3 Responder Rate

To evaluate the persistent antimicrobial properties of a single Swabstick impregnated with 2% (w/v) chlorhexidine gluconate in 70% (v/v) isopropyl alcohol,  $\log_{10}$  bacterial counts at 6 hours post-product application for each product application site will be converted to a binary (yes or no) success measure with success defined as having skin flora counts that are less than or equal to the baseline skin flora counts.



#### 6.1.4 Product Weight

The weight (grams) of product solutions applied to an anatomical area will be estimated as:

Product weight prior to product application (g) - product weight post-product application (g)

#### 6.2 Analysis Methods

#### 6.2.1 HC Analysis

#### 6.2.1.1 Summary Statistics

The following descriptive statistics for  $\log_{10}$  CFU/cm<sup>2</sup> at each time point (baseline, 30 seconds, 10 minutes and 6 hours) and  $\log_{10}$  CFU/cm<sup>2</sup> reductions at each post application sampling time point (30 seconds, 10 minutes and 6 hours) will be computed for the IP and RS, grouped by anatomical site: mean, median, standard deviation, minimum, maximum, and count (cf. Tables A.2.1 and A.2.2).

#### 6.2.1.2 Primary Analysis

The 95% confidence intervals (two-sided) will be calculated for the average log reductions for the IP and RS at each post application sampling time point on each anatomical area using one-sample t-test (two-sided). The 95% confidence lower bound for mean log reduction at 30 seconds and 6 hours will be compared to the acceptance criteria (cf. Table A.2.4).

- If the lower limit of the 95% confidence interval (two-sided) of mean log reduction at 30 seconds is greater than or equal to 2 on the abdomen, acceptance criteria are met on the abdomen at 30 seconds.
- If the lower limit of the 95% confidence interval (two-sided) of mean log reduction at 30 seconds is greater than or equal to 3 on the groin, acceptance criteria are met on the groin at 30 seconds.
- If the lower limit of the 95% confidence interval (two-sided) of mean log reduction at 6 hours is greater than or equal to 2 on the abdomen, acceptance criteria are met on the abdomen at 6 hours.
- If the lower limit of the 95% confidence interval (two-sided) of mean log reduction at 6 hours is greater than or equal to 3 on the groin, acceptance criteria are met on the groin at 6 hours.

The RS will be also compared to the acceptance criteria applied to the IP.

#### 6.2.1.3 Exploratory Analysis

The same analysis as described in Section 6.2.1.2 will be performed for log reduction at the 10 minute time point on each anatomical area for the IP and RS using one-sample t-test (two-sided) (cf. Table A.2.5).

Log<sub>10</sub> CFU/cm<sup>2</sup> reductions at 30 seconds, 10 minutes, and 6 hours on the abdomen and the groin for the IP will be compared to the RS using two-sample t-test (two-sided). Difference in log reduction along with 95% confidence interval (CI) at each post application sampling time point will be compared to zero. If 95% CI contains zero, the conclusion is no significant difference in log reduction between IP and RS. If 95% CI does not contain zero, the conclusion is significant difference in log reduction exists and the direction of the difference will be indicated (cf. Table A.2.6).



A graph for the log reduction at each post application sampling time point with 95% confidence interval will be provided (cf. Figure C.1.1 created based on the simulated data).

#### 6.2.2 FDA Analysis

#### 6.2.2.1 Summary Statistics

The following descriptive statistics for  $\log_{10} \text{ CFU/cm}^2$  at each time point (baseline, 30 seconds, 10 minutes and 6 hours) and  $\log_{10} \text{ CFU/cm}^2$  reductions at each post application sampling time point (30 seconds, 10 minutes and 6 hours) will be computed for the IP, AC and NC, grouped by anatomical site: mean, median, standard deviation, minimum, maximum, and count (cf. Tables A.3.1 and A.3.2).

Responder rates at 6 hours post-product application will be summarized descriptively for each product (IP, AC and NC) on each body site. No inferential analysis will be performed on the responder rates at 6 hours post-product application (cf. Table A.3.3).

The following descriptive statistics for product weight will be computed for the IP, AC and NC, grouped by anatomical site: mean, median, standard deviation, minimum, maximum, and count (cf. Table A.3.4).

#### 6.2.2.2 Primary Analysis

A linear regression model for each body site (abdomen or groin) will be used for primary analysis of efficacy at 10 minutes. In the model, the response is the post-product application bacterial counts at 10 minutes and predictors are the study products (IP, AC or NC) as a fixed effect and the preproduct application bacterial loads as a covariate. The average treatment effect (ATE) corrected for pre-product application bacterial loads will be estimated from the model and compared to both non-inferiority and superiority criteria (cf. Table A.3.5).

For assessment of the four primary objectives (i.e., immediate activity at 10 minutes post application on the abdomen and groin for non-inferiority and superiority):

- A non-inferiority criterion with a 0.5 log<sub>10</sub> margin will be implemented for ATE of the IP compared to the AC (i.e., if the upper two-sided 95% confidence bound of the post-product application bacterial load corrected for pre-product application bacterial load of the IP-AC is less than 0.5 log<sub>10</sub>, the non-inferiority criterion is met).
- A 1.2 log<sub>10</sub> superiority criterion will be implemented for the ATE of the IP compared to the NC (i.e., if the lower two-sided 95% confidence bound of the post-product application bacterial load corrected for pre-product application bacterial load of the NC-IP is greater than 1.2 log<sub>10</sub>, the superiority criterion is met).

A graph showing the ATE with 95% confidence intervals for post-product log CFU at 10 minutes correcting for pre-product application will be provided for each contrast (cf. Figure C.2.1 created based on the simulated data).

#### 6.2.2.3 Secondary Analysis

A gatekeeping procedure will be applied: the efficacy analysis for two secondary objectives [30-second (abdomen only) post-product application time point] will be performed only when all four primary



objectives [10-minute (abdomen and groin) post-product application time point] pass the acceptance criteria.

A linear regression model for abdomen only will be used for secondary analysis of efficacy at 30 seconds. In the model, the response is the post-product application bacterial counts at 30 seconds and predictors are the study products (IP, AC or NC) as a fixed effect and the pre-product application bacterial loads as a covariate. The average treatment effect (ATE) corrected for pre-product application bacterial loads will be estimated from the model and compared to both non-inferiority and superiority criteria (cf. Table A.3.6).

For assessment of the two secondary objectives (i.e., immediate activity at 30 seconds post application on the abdomen for non-inferiority and superiority):

- A non-inferiority criterion with a 0.5 log<sub>10</sub> margin will be implemented for ATE of the IP compared to the AC (i.e., if the upper two-sided 95% confidence bound of the post-product application bacterial load corrected for pre-product application bacterial load of the IP-AC is less than 0.5 log<sub>10</sub>, the non-inferiority criterion is met).
- A 1.2 log<sub>10</sub> superiority criterion will be implemented for the ATE of the IP compared to the NC (i.e., if the lower two-sided 95% confidence bound of the post-product application bacterial load corrected for pre-product application bacterial load of the NC-IP is greater than 1.2 log<sub>10</sub>, the superiority criterion is met).

A graph showing the ATE with 95% confidence intervals for post-product log CFU at 30 seconds correcting for pre-product application will be provided for each contrast if acceptance criteria are met for all four co-primary objectives (cf. Figure C.2.1 created based on the simulated data). If acceptance criteria are not met for any of four co-primary objectives, the plot for 30 seconds will be removed from the graph as no analysis for 30 seconds is performed.

#### 6.2.3 Safety Analysis

Skin irritation scores for each product at each post application sampling time per body location will be tabulated with frequency and percentage (cf. Table A.4.1) for ITT population set (all randomized subjects that received study product).

The statistical significance of differences in skin irritation between the study products at each post application sampling time will be evaluated by Fisher's exact test on skin irritation data summarized for safety analysis as follows: any reaction above a zero (no reaction) on the skin irritation rating scale for any category (erythema, edema, rash, and dryness) will be considered a positive signal for that substance (cf. Table A.4.3). If Fisher's exact test shows statistically significant skin irritation between the study products, follow-up analyses (e.g., Fisher's exact test for subgroup analysis) may be conducted to determine how the reactions differ (cf. Table A.4.4).

Adverse events (AEs) will be listed for all enrolled subjects (cf. Listing B.6). Whether subjects are in ITT population set (randomized subjects that received study product) will be indicated. A summary showing number and percentage of subjects with AE(s) observed will be provided for ITT population set (cf. Table A.4.2). No inferential analysis will be performed on the incidence of AEs. If any serious adverse events (SAEs) happen, more details for SAEs will be listed (cf. Listing B.7).



#### 6.3 Adjustments for Multiple Objectives

An overall significance level of 0.05 ( $\alpha = 0.05$ ) is used.

This study has two sets of objectives, one for Health Canada (HC) analysis and the other for US FDA analysis. These two sets of objectives are considered independently of each other and no multiplicity adjustment between two sets of objectives is performed.

Within the HC analysis primary objectives, since the study HC efficacy analysis will declare success when and only when all four primary objectives pass HC analysis acceptance criteria, no multiplicity adjustment is required [3].

Within the FDA efficacy analysis, a gatekeeping procedure will be applied: the efficacy analysis for two secondary objectives [30-second (abdomen only) post-product application time point] will be performed only when all four primary objectives [10-minute (abdomen and groin) post-product application time point] pass the acceptance criteria. No multiplicity adjustment between primary and secondary objectives is performed. For primary objectives [10-minute (abdomen and groin) post-product application time point], since it will declare success when and only when all four primary objectives pass FDA analysis acceptance criteria, no multiplicity adjustment for the four primary objectives is required [3]. For secondary objectives [30-second (abdomen only) post-product application time point], since it will declare success when and only when all four primary and two secondary objectives pass FDA analysis acceptance criteria, no multiplicity adjustment for the two secondary objectives is required [3].

#### 6.4 Handling of Missing Data and Sensitivity Analysis

Missing log<sub>10</sub> CFU/cm<sup>2</sup> determinations at 30 seconds, 10 minutes, or 6 hours, such as due to laboratory error or subject lost to follow up, will be reported as missing and will not be imputed for main analyses (log reduction, ATE and responder rate) as described in Section 6.2. Missing product weight will be also reported as missing and will not be imputed. Details of any missing data and rationale for inclusion/exclusion in the mITT or PP data set will be described in the statistical or study report.

Sensitivity analysis will be performed to evaluate the impact of missing data, if any, for primary and secondary objectives (refer to Section 6.4.1 for details).

- For HC analysis (log reduction), if acceptance criteria are met for primary objectives, sensitivity analysis will be performed for primary objectives based on the mITT population sets. No sensitivity analysis will be performed if acceptance criteria are not met for primary objectives.
- For FDA analysis (ATE), if acceptance criteria are met for both primary and secondary objectives, sensitivity analysis will be performed separately for primary and secondary objectives based on the mITT population sets. If acceptance criteria are met for primary objectives but not for secondary objectives, sensitivity analysis will be only performed for primary objectives based on the mITT population sets and no sensitivity analysis will be performed for secondary objectives. No sensitivity analysis will be performed if acceptance criteria are not met for primary objectives.
- No sensitivity analysis will be performed for exploratory objectives.



#### 6.4.1 Sensitivity Analysis

For  $\log_{10}$  CFU/cm<sup>2</sup> determinations, multiple imputation under the assumption that data are missing at random (MAR) will be performed to impute a series of  $\log_{10}$  CFU values relative to the baseline  $\log_{10}$  CFU values for all missing data points.

- For HC objectives, the multiple imputation will be performed separately for each of the four primary objectives (IP only).
- For FDA objectives, the multiple imputation will be performed separately for each of the four primary and two secondary objectives.

If results based on imputed data meet the acceptance criteria, a tipping-point sensitivity analysis will be performed by shifting the imputed values to assess how severe departures from missing at random (MAR) must be in order to find the tipping point at which the acceptance criteria would not be met.

Multiple imputation and tipping point approaches for either HC objectives or FDA objectives include the following steps:

- 1. The missing data are filled in 25 times to generate 25 complete data sets using Predictive Mean Matching (PPM) method provided in R package "MICE".
- 2. Each of the 25 complete data sets are analyzed by using routine analysis method applied for log reduction analysis (HC objectives) or for ATE analysis (FDA objectives).
- 3. The results from the 25 complete data sets are combined/pooled for the inference and compared to the acceptance criteria (cf. Tables A.5.1 for HC objectives and A.5.2 for FDA objectives).
- 4. If results based on imputed data meet the acceptance criteria, repeat Step 1 to generate multiple imputed data sets, with a specified shift parameter that shifts the imputed values (shift parameter will be applied to the IP group only).
  - For log reduction, the shift parameter will start from -0.1 to smaller (more stringent) numbers (i.e., -0.1, -0.2, ...).
  - For ATE of IP-AC or NC-IP, the shift parameter will start from 0.1 to larger (more stringent) numbers (i.e., 0.1, 0.2, ...);
- 5. Repeat Step 2 for the imputed data sets with shift parameter applied.
- 6. Repeat Step 3 to obtain the estimate and 95% confidence limits to see if acceptance criteria are met.
- 7. Repeat Steps 4-6 with more stringent shift parameters applied until acceptance criteria are not met.

The tipping point for the shift parameter that reverses the conclusion ("Met Criteria" changes from "Yes" to "No") will be listed (cf. Tables A.5.3 for HC objectives and A.5.4 for FDA objectives).

For responder rate at 6 hours (FDA objectives), subjects with missing  $\log_{10}$  CFU/cm<sup>2</sup> determinations at 6 hours will not be excluded from sensitivity analysis. Missing data will be imputed by increasing the assumed number of failures sequentially from 0/M to M/M, where M is the number of missing data points at 6 hours. This sensitivity analysis will be performed for all products (IP, AC and NC) on each anatomical site and will provide information on the possible effect of missing data on study results (cf. Table A.5.5).



#### 6.5 Demographics/Other Descriptive Information

Demographics: Table A.6.1 shows demographics information for subjects in ITT population sets.

Procedure Overview: Any sampling fluid from sampling site that extended to other remaining sites at a certain time point will be listed for each body location (cf. Listing B.8). Any dressing application that was placed on the application site at the 10-minute time point and dressing integrity was compromised any time prior to the 6-hour time point will be listed for each body location (cf. Listing B.9). This will be based on data from ITT population sets.

Core Lab Overview: Any sampling solution that was lost at any time during the procedure will be listed with time points affected (cf. Listing B.10). This will be based on data from ITT population sets.

Product Failures/Lab Accidents/User Errors: Any product failures/lab accidents/user errors will be listed for all study products used (cf. Listing B.11).



### 7 References

- [1] ASTM E1173-15. Standard Test Method for Evaluation of Preoperative, Precatheterization, or Preinjection Skin Preparations. ASTM International, West Conshohocken, PA, 2015.
- [2] R Core Team. R: A Language and Environment for Statistical Computing. R Foundation for Statistical Computing, Vienna, Austria, 2016. URL https://www.R-project.org/.
- [3] Frank Bretz. Alex Dmitrienko, Ajit C.Tamhane. Multiple Testing Problems in Pharmaceutical Statistics. Chapman and Hall/CRC, 2009.



## 8 Appendix

### A Tables

### A.1 Analysis Population Set(s)

Table A.1.1: Overall Subject Disposition

| Number of Subjects | Comments |
|--------------------|-----------------------|
| n | |
| n | |
| n | |
| n | |
| n | |
| n | |
| | n<br>n<br>n<br>n<br>n |

Table A.1.2: Number of Evaluable Subjects for HC Analysis

| Body Location | Population Sets | IP | RS | Overall |
|---------------|---------------------------|--------------|----|--------------|
| Abdomen/Groin | ITT Safety | n | n | n |
| | mITT CFU Count 30 Seconds | $\mathbf{n}$ | n | n |
| | PP CFU Count 30 Seconds | $\mathbf{n}$ | n | $\mathbf{n}$ |
| | mITT CFU Count 10 Minutes | $\mathbf{n}$ | n | n |
| | PP CFU Count 10 Minutes | n | n | n |
| | mITT CFU Count 6 Hours | n | n | n |
| | PP CFU Count 6 Hours | $\mathbf{n}$ | n | $\mathbf{n}$ |
| | mITT Product Weight | n | n | n |
| | PP Product Weight | n | n | n |

Table A.1.3: Number of Evaluable Subjects for FDA Analysis

| | | · · | | · · | |
|---|---|---|---|---|---|
| Body Location | Population Sets | IP | AC | NC | Overall |
| Abdomen/Groin | ITT Safety | n | n | n | n |
| | mITT CFU Count 30 Seconds | $\mathbf{n}$ | $\mathbf{n}$ | n | $\mathbf{n}$ |
| | PP CFU Count 30 Seconds | $\mathbf{n}$ | $\mathbf{n}$ | n | $\mathbf{n}$ |
| | mITT CFU Count 10 Minutes | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ |
| | PP CFU Count 10 Minutes | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ |
| | mITT Responder Rate 6 Hours | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ |
| | PP Responder Rate 6 Hours | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ |
| | mITT Product Weight | $\mathbf{n}$ | $\mathbf{n}$ | n | n |
| | PP Product Weight | $\mathbf{n}$ | $\mathbf{n}$ | n | n |



### A.2 HC Analysis

Table A.2.1: mITT/PP - Summary Statistics for HC Analysis - Log CFU

| | | 7 | | | 0 | | |
|---|---|---|---|---|---|---|---|
| Body Location | Product | Time Point | Count | Mean | Median | $\operatorname{SD}$ | Range |
| | | | | | | | (Min-Max) |
| Abdomen/Groin | IP/RS | Baseline | n | X.XX | x.xx | X.XX | x.xx - x.xx |
| | | 30 Seconds | $\mathbf{n}$ | X.XX | X.XX | X.XX | x.xx - x.xx |
| | | 10 Minutes | $\mathbf{n}$ | X.XX | X.XX | X.XX | x.xx - x.xx |
| | | 6 Hours | n | X.XX | x.xx | X.XX | x.xx - x.xx |

Table A.2.2: mITT/PP - Summary Statistics for HC Analysis - Log Reduction

| | , | • | | · | | | |
|---|---|---|---|---|---|---|---|
| Body Location | Product | Time Point | Count | Mean | Median | SD | Range |
| | | | | | | | (Min-Max) |
| Abdomen/Groin | IP/RS | 30 Seconds | n | X.XX | x.xx | X.XX | X.XX - X.XX |
| | | 10 Minutes | $\mathbf{n}$ | X.XX | X.XX | X.XX | X.XX - X.XX |
| | | 6 Hours | n | X.XX | x.xx | X.XX | x.xx - x.xx |

Table A.2.3: mITT/PP - Summary Statistics for HC Analysis - Product Weight

| Body Location | Product | Count | Mean | Median | SD | Range<br>(Min-Max) |
|---------------|---------|-------|------|--------|------|--------------------|
| Abdomen/Groin | IP/RS | n | x.xx | x.xx | X.XX | x.xx - x.xx |

Table A.2.4: mITT/PP - Analysis Results for HC Analysis - Log Reduction at 30 Seconds and 6 Hours

| Body Location | Product | Time Point | Count | Mean Log Reduction (95% CI) | Met Criteria |
|---|---|---|---|---|---|
| Abdomen/Groin | IP/RS | 30 Seconds | n | x.xx (x.xx, x.xx) | Yes/No |
| | | 6 Hours | n | x.xx(x.xx, x.xx) | Yes/No |



Table A.2.5: mITT/PP - Analysis Results for for HC Analysis - Log Reduction at 10 Minutes

| Body Location | Product | Time Point | Count | Mean Log Reduction (95% CI) |
|---------------|---------|------------|-------|-----------------------------|
| Abdomen/Groin | IP/RS | 10 Minutes | n | x.xx (x.xx, x.xx) |

Table A.2.6: mITT/PP - Analysis Results for for HC Analysis - Difference in Log Reduction

| | / | <i>J</i> | | 0 |
|---|---|---|---|---|
| Body Location | Contrast | Time Point | Difference in Log Reduction | Conclusion |
| | | | (95% CI) | |
| Abdomen/Groin | IP-RS | 30 Seconds | x.xx (x.xx, x.xx) | Sign. Diff/No Sign. Diff |
| Abdomen/Groin | IP-RS | 10 Minutes | x.xx(x.xx, x.xx) | Sign. Diff/No Sign. Diff |
| Abdomen/Groin | IP-RS | 6 Hours | x.xx(x.xx, x.xx) | Sign. Diff/No Sign. Diff |



### A.3 FDA Analysis

Table A.3.1: mITT/PP - Summary Statistics for FDA Analysis - Log CFU

| | | • | | | | | |
|---|---|---|---|---|---|---|---|
| Body Location | Product | Time Point | Count | Mean | Median | $^{\mathrm{SD}}$ | Range |
| | | | | | | | (Min-Max) |
| Abdomen/Groin | IP/AC/NC | Baseline | n | x.xx | x.xx | x.xx | x.xx - x.xx |
| | | 30 Seconds | n | X.XX | x.xx | X.XX | X.XX - X.XX |
| | | 10 Minutes | n | X.XX | x.xx | X.XX | X.XX - X.XX |
| | | 6 Hours | n | x.xx | x.xx | x.xx | x.xx - x.xx |

Table A.3.2: mITT/PP - Summary Statistics for FDA Analysis - Log Reduction

| Body Location | Product | Time Point | Count | Mean | Median | SD | Range<br>(Min-Max) |
|---|---|---|---|---|---|---|---|
| Abdomen/Groin | IP/AC/NC | 30 Seconds | n | x.xx | x.xx | X.XX | x.xx - x.xx |
| | | 10 Minutes | n | x.xx | x.xx | x.xx | x.xx - x.xx |
| | | 6 Hours | n | x.xx | x.xx | X.XX | x.xx - x.xx |
| | | 6 Hours | n | x.xx | X.XX | X.XX | _ |

Table A.3.3: mITT/PP - Summary Statistics for FDA Analysis - Responder Rate at 6 Hours

| Body Location | Product | Responder Rate |
|---------------|----------|----------------|
| Abdomen/Groin | IP/AC/NC | n/N (%) |

Note: n is number of responders and N is total number of evaluable subjects.

Table A.3.4: mITT/PP - Summary Statistics for FDA Analysis - Product Weight

| | / | J .= | | | | |
|---------------|----------|-------|------|--------|------|-------------|
| Body Location | Product | Count | Mean | Median | SD | Range |
| | | | | | | (Min-Max) |
| Abdomen/Groin | IP/AC/NC | n | x.xx | X.XX | x.xx | x.xx - x.xx |



Table A.3.5: mITT/PP - Analysis Results for FDA Analysis - ATE at 10 Minutes

| Body Location | Contrast | Time Point | ATE (95% CI) | Met Criteria |
|---------------|----------|------------|-------------------|--------------|
| Abdomen/Groin | IP-AC | 10 Minutes | x.xx (x.xx, x.xx) | Yes/No |
| Abdomen/Groin | NC-IP | 10 Minutes | x.xx (x.xx, x.xx) | Yes/No |

Table A.3.6: mITT/PP - Analysis Results for for FDA Analysis - ATE at 30 Seconds

| Body Location | Contrast | Time Point | ATE (95% CI) | Met Criteria |
|---------------|----------|------------|-------------------|--------------|
| Abdomen | IP-AC | 30 Seconds | x.xx (x.xx, x.xx) | Yes/No |
| Abdomen | NC-IP | 30 Seconds | x.xx(x.xx, x.xx) | Yes/No |



### A.4 Safety Analysis

Table A.4.1: ITT - Summary Statistics for Irritation Scores for Abdomen/Groin at Baseline/30 Seconds/10 Minutes/6 Hours

| Characteristic | IP | RS | AC | NC | Overall |
|----------------------------------|-------|-------|-------|-------|---------|
| Erythema | | | | | |
| 0-No reaction | n (%) | n (%) | n (%) | n (%) | n (%) |
| 1-Mild and/or transient redness | n (%) | n (%) | n (%) | n (%) | n (%) |
| 2-Moderate redness | n (%) | n (%) | n (%) | n (%) | n (%) |
| 3-Severe redness | n (%) | n (%) | n (%) | n (%) | n (%) |
| Edema | | | | | |
| 0-No reaction | n (%) | n (%) | n (%) | n (%) | n (%) |
| 1-Mild and/or transient swelling | n (%) | n (%) | n (%) | n (%) | n (%) |
| 2-Moderate swelling | n (%) | n (%) | n (%) | n (%) | n (%) |
| 3-Severe swelling | n (%) | n (%) | n (%) | n (%) | n (%) |
| Rash | | | | | |
| 0-No reaction | n (%) | n (%) | n (%) | n (%) | n (%) |
| 1-Mild and/or transient rash | n (%) | n (%) | n (%) | n (%) | n (%) |
| 2-Moderate rash | n (%) | n (%) | n (%) | n (%) | n (%) |
| 3-Severe rash | n (%) | n (%) | n (%) | n (%) | n (%) |
| Dryness | | | | | |
| 0-No reaction | n (%) | n (%) | n (%) | n (%) | n (%) |
| 1-Mild and/or transient dryness | n (%) | n (%) | n (%) | n (%) | n (%) |
| 2-Moderate dryness | n (%) | n (%) | n (%) | n (%) | n (%) |
| 3-Severe dryness | n (%) | n (%) | n (%) | n (%) | n (%) |

Table A.4.2: ITT - Adverse Events Summary

| Characteristic | IP | RS | AC | NC | Overall |
|----------------|-------|-------|-------|-------|---------|
| Adverse Events | | | | | |
| No | n (%) | n (%) | n (%) | n (%) | n (%) |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) |

Note: Overall column is calculated based on overall unique subjects included in ITT.



Table A.4.3: ITT - Safety Analysis - Overall Comparisons for Erythema/Edema/Rash/Dryness

| Body Location | Time Point | p-value | Conclusion |
|---------------|------------|---------|--------------------------|
| Abdomen/Groin | 30 Seconds | 0.xxx | Sign. Diff/No Sign. Diff |
| Abdomen/Groin | 10 Minutes | 0.xxx | Sign. Diff/No Sign. Diff |
| Abdomen/Groin | 6 Hours | 0.xxx | Sign. Diff/No Sign. Diff |

Note: If analysis is not applicable, p-value will be shown as "N/A".

Table A.4.4: ITT - Safety Analysis - Subgroup Comparisons for Irritation Scores

| | | v | J | 0 1 | 1 | |
|---|---|---|---|---|---|---|
| _ | Body Location | Characteristic | Time | Compar- | Odds Ratio (95% | Conclusion |
| | | | Point | ison | CI) | |
| - | Abdomen/Groin | | | | x.xx (x.xx, x.xx) | Sign. Diff/No Sign. Diff |



### A.5 Sensitivity Analysis

Table A.5.1: Pooled Analysis Results Based on Imputated Datasets for HC Objectives - Log Reduction

| | · | • | | • |
|---------------|---------|------------|-------------------|--------------|
| Body Location | Product | Time Point | Log Reduction | Met Criteria |
| | | | (95% CI) | |
| Abdomen/Groin | IP | 30 Seconds | x.xx (x.xx, x.xx) | Yes/No |
| | IP | 6 Hours | x.xx(x.xx, x.xx) | Yes/No |

Table A.5.2: Pooled Analysis Results Based on Imputated Datasets for FDA Objectives - ATE

| Body Location | Time Point | Contrast | ATE (95% CI) | Met Criteria |
|---------------|------------|----------|-------------------|--------------|
| Abdomen/Groin | 10 Minutes | IP-AC | x.xx (x.xx, x.xx) | Yes/No |
| | 10 Minutes | NC-IP | x.xx (x.xx, x.xx) | Yes/No |
| Abdomen | 30 Seconds | IP-AC | x.xx (x.xx, x.xx) | Yes/No |
| | 30 Seconds | NC-IP | x.xx (x.xx, x.xx) | Yes/No |

Table A.5.3: Tipping Point Analysis for HC Objectives - Log Reduction

| | • | · | _ | |
|---|---|---|---|---|
| Product | Time Point | Shift | Log Reduction | Met Criteria |
| | | Parameter | (95% CI) | |
| IP | 30 Seconds | -X.X | x.xx (x.xx, x.xx) | Yes |
| IP | 30 Seconds | -X.X | x.xx(x.xx, x.xx) | Yes |
| IP | 30 Seconds | -x.x | x.xx(x.xx, x.xx) | No |
| IP | 6 Hours | -X.X | x.xx(x.xx, x.xx) | Yes |
| IP | 6 Hours | -X.X | x.xx(x.xx, x.xx) | Yes |
| IP | 6 Hours | -x.x | x.xx (x.xx, x.xx) | No |
| | IP<br>IP<br>IP<br>IP<br>IP | IP 30 Seconds IP 30 Seconds IP 30 Seconds IP 6 Hours IP 6 Hours | IP 30 Seconds -x.x IP 30 Seconds -x.x IP 30 Seconds -x.x IP 6 Hours -x.x IP 6 Hours -x.x IP 6 Hours -x.x | IP 30 Seconds -x.x x.xx (x.xx, x.xx) IP 30 Seconds -x.x x.xx (x.xx, x.xx) IP 30 Seconds -x.x x.xx (x.xx, x.xx) IP 6 Hours -x.x x.xx (x.xx, x.xx) IP 6 Hours -x.x x.xx (x.xx, x.xx) IP 6 Hours -x.x x.xx (x.xx, x.xx) |



Table A.5.4: Tipping Point Analysis for FDA Objectives - ATE

| | 1.1 | O v | · · | | |
|---|---|---|---|---|---|
| Body Location | Time Point | Contrast | Shift | ATE (95% CI) | Met Criteria |
| | | | Parameter | | |
| Abdomen/Groin | 10 Minutes | IP-AC | X.X | x.xx (x.xx, x.xx) | Yes |
| | 10 Minutes | IP-AC | X.X | x.xx(x.xx, x.xx) | Yes |
| | 10 Minutes | IP-AC | X.X | x.xx(x.xx, x.xx) | No |
| | 10 Minutes | NC-IP | X.X | x.xx(x.xx, x.xx) | Yes |
| | 10 Minutes | NC-IP | X.X | x.xx(x.xx, x.xx) | Yes |
| | 10 Minutes | NC-IP | X.X | x.xx(x.xx, x.xx) | No |
| Abdomen | 30 Seconds | IP-AC | X.X | x.xx (x.xx, x.xx) | Yes |
| | 30 Seconds | IP-AC | X.X | x.xx(x.xx, x.xx) | Yes |
| | 30 Seconds | IP-AC | X.X | x.xx(x.xx, x.xx) | No |
| | 30 Seconds | NC-IP | X.X | x.xx(x.xx, x.xx) | Yes |
| | 30 Seconds | NC-IP | X.X | x.xx(x.xx, x.xx) | Yes |
| | 30 Seconds | NC-IP | X.X | x.xx(x.xx, x.xx) | No |
| • | · | | · | · | |

Table A.5.5: Sensitivity Analysis for FDA Objectives - Responder Rate at 6 Hours

| Body Location | Product | Subjects Imputed to Non-responders | Responder Rate |
|---|---|---|---|
| Abdomen/Groin | IP/AC/NC | +0 | n/N (%) |
| | | +1 | n/N (%) |
| | | +2 | n/N (%) |
| | | | n/N (%) |
| | | +M | n/N (%) |

Note: Subjects imputated to non-responders are added to the denominator (N) for the responder rate.



### A.6 Demographics

Table A.6.1: ITT - Demographics

| | | • | | | |
|---|---|---|---|---|---|
| Characteristic | IP | RS | AC | NC | Overall |
| Age at Time of Informed Consent (Years) | | | | | |
| Mean | X.X | X.X | X.X | X.X | X.X |
| Median | X.X | X.X | x.x | X.X | x.x |
| $\operatorname{SD}$ | X.X | X.X | X.X | X.X | x.x |
| Min, Max | X.X | X.X | X.X | X.X | x.x |
| Total Count | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ | $\mathbf{n}$ |
| Gender | | | | | |
| Male | n (%) | n (%) | n (%) | n (%) | n (%) |
| Female | n (%) | n (%) | n (%) | n (%) | n (%) |
| Ethnicity | | | | | |
| Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) |
| Not Hispanic or Latino | n (%) | n (%) | n (%) | n (%) | n (%) |
| Race | | | | | |
| American Indian or Alaska Native | n (%) | n (%) | n (%) | n (%) | n (%) |
| Asian | n (%) | n (%) | n (%) | n (%) | n (%) |
| Black or African American | n (%) | n (%) | n (%) | n (%) | n (%) |
| Native Hawaiian or Other Pacific Islander | n (%) | n (%) | n (%) | n (%) | n (%) |
| White | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) |
| N-4 O111 :11-41 h1 | . , | | ` ' | ` ' | \ / |

Note: Overall column is calculated based on overall unique subjects included in ITT.



# B Listings

Table B.1: Protocol Deviations

| RandID | Nature of Deviation | Additional Details |
|--------|---------------------|--------------------|
| Rxxxx | | |
| Rxxxx | | |
| Rxxxx | | |
| Rxxxx | | |

Table B.2: Subjects with Excluded Data for HC Analysis

| RandID | Body | Product | Time Point | Included in | Included in |
|--------|----------|---------|------------|-------------|-------------|
| | Location | | | mITT CFU | PP CFU |
| | | | | Count | Count |
| Rxxxx | | | | Yes/No | Yes/No |
| Rxxxx | | | | Yes/No | Yes/No |
| Rxxxx | | | | Yes/No | Yes/No |
| Rxxxx | | | | Yes/No | Yes/No |

Table B.3: Subjects with Excluded Data for FDA Analysis

| | | | · · | | | | · | | |
|---|---|---|---|---|---|---|---|---|---|
| RandID | Body | Product | Time | Included | Included | Included | Included | Included | Included |
| | Location | | Point | in $mITT$ | in PP | in mITT | in PP | in $mITT$ | in PP |
| | | | | CFU | CFU | Responder | Responder | Product | Product |
| | | | | Count | Count | Rate | Rate | Weight | Weight |
| Rxxxx | | | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No |

Table B.4: Subjects who Did Not Complete the Study

| RandID | Subject's Status | Comments |
|--------|------------------|----------|
| Rxxxx | Screen Failure | |
| Rxxxx | | |
| Rxxxx | | |
| Rxxxx | | |



Table B.5: Subjects Not Passing Treatment-day Baseline Criteria

| RandID | Body Location | Product | Time Point | Result $(\log_{10})$ |
|--------|---------------|---------|------------|----------------------|
| Rxxxx | | | | X.XX |
| Rxxxx | | | | X.XX |
| Rxxxx | | | | X.XX |
| Rxxxx | | | | X.XX |

#### Table B.6: Adverse Events

| Ran-<br>dID | AE<br>Term | Start Date | End Date | AE<br>Out-<br>come | Severity | Relation-<br>ship to<br>Device | Relation-<br>ship to<br>Procedure | SAE | Additional<br>Details | In-<br>cluded<br>in<br>ITT |
|---|---|---|---|---|---|---|---|---|---|---|
| Rxxxx | | | | | | | | Yes/No | | Yes/No |
| Rxxxx | | | | | | | | Yes/No | | Yes/No |
| Rxxxx | | | | | | | | Yes/No | | Yes/No |
| Rxxxx | | | | | | | | Yes/No | | Yes/No |

### Table B.7: Serious Adverse Events

| RandID | AE Term | Start Date | End Date | Serious | Hospital | Hospital | Was SAE Unex- | Included |
|---|---|---|---|---|---|---|---|---|
| | | | | Criteria | Admission | Discharge | pected/Unanticipa | ted in ITT |
| | | | | | Date | Date | | |
| Rxxxx | | | | | | | Yes/No | Yes/No |
| Rxxxx | | | | | | | Yes/No | Yes/No |
| Rxxxx | | | | | | | Yes/No | Yes/No |
| Rxxxx | | | | | | | Yes/No | Yes/No |

### Table B.8: Procedure Overview - Sampling Fluid

| RandID | D Body Location Product | | Did Sampling Fluid<br>from Sampling Site | Time Points Affected |
|---|---|---|---|---|
| | | Extend to Other | | |
| | | | Remaining Sites at | |
| | | | Any Time Point | |
| Rxxxx | | | Yes | 30 Seconds |
| Rxxxx | | | Yes | |
| Rxxxx | | | Yes | |
| Rxxxx | | | Yes | |



Table B.9: Procedure Overview - Dressing Application

| RandID | Body | Product | Was Dressing | Was Dressing | Details |
|---|---|---|---|---|---|
| | Location | | Application Placed | Integrity | |
| | | | on the Application | Compromised at Any | |
| | | | Site at the 10 Minute | Time Prior to the 6 | |
| | | | Time Point | Hour Time Point | |
| Rxxxx | | | Yes | Yes | Subject Confirmed |
| | | | | | Dressing was |
| | | | | | Adjusted and/or |
| | | | | | Touched |
| Rxxxx | | | Yes | Yes | |
| Rxxxx | | | Yes | Yes | |
| Rxxxx | | | Yes | Yes | |

Table B.10: Core Lab Procedure Overview - Sample Solution

| RandID | Body | Product | Was Any Sampling | Time Point Affected | Volume Remaining |
|---|---|---|---|---|---|
| | Location | | Solution Lost at Any | | (mL) |
| | | | Time During the | | |
| | | | Procedure | | |
| Rxxxx | | | Yes | Baseline | |
| Rxxxx | | | Yes | | |
| Rxxxx | | | Yes | | |
| Rxxxx | | | Yes | | |

Table B.11: Product Failures/Lab Accidents/User Errors

| RandID | Are There Any | Date of | Product | Time of | Incident | Details | Was | Was an |
|---|---|---|---|---|---|---|---|---|
| | Product | Incident | Affected | Incident | $\operatorname{Code}$ | | Product | AE |
| | Failures/Lab | | | | | | Used on | Associated |
| | Accidents/User | | | | | | Study | with the |
| | Errors to Report | | | | | | Subject | Incident |
| Rxxxx | Yes | | | During | Product | | | |
| | | | | Product | Handling | | | |
| | | | | Exposure | Issue | | | |
| Rxxxx | Yes | | | | | | | |
| Rxxxx | Yes | | | | | | | |
| Rxxxx | Yes | | | | | | | |



# C Figures

## C.1 HC Analysis



Figure C.1.1: mITT/PP - Log Reduction with 95% CI (Example Data Only)



### C.2 FDA Analysis



Figure C.2.1: mITT/PP - ATE with 95% CI (Example Data Only)